CLINICAL TRIAL: NCT03676179
Title: The Comparison of Anterior Knee Pain in Patella With or Without Denervation in Medial Unicompartmental Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Pranungkraw General Hospital (Unknown)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, principle investigator, Ramathibodi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08/2561
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: unicompartment knee arthroplasty with patella denervation
Who Masked: Investigator, Outcomes Assessor
Masking Description: unicompartment knee arthroplasty without patella denervation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unicompartment knee arthroplasty and patella denervation (Active Comparator): UKA and patella denervation
  Interventions: Procedure: patella denervation
- unicompartment knee arthroplasty and patella non-denervation (Experimental): UKA and patella non-denervation
  Interventions: Procedure: patella non-denervation

INTERVENTIONS:
Procedure: patella denervation — patella denervation
  Arms: unicompartment knee arthroplasty and patella denervation
Procedure: patella non-denervation — patella non-denervation
  Arms: unicompartment knee arthroplasty and patella non-denervation

SUMMARY:
the present study will conduct to assess anterior knee pain and complications after medial UKA with or without patella denervation in medial compartment arthritis and severe lateral facet patellofemoral arthritis patients.

DETAILED DESCRIPTION:
In this prospective cohort study, the investigators will conduct to compare the clinical result of 70 patients of unicompartment knee arthroplasty with and without patella denervation between April, 2018 and April, 2019 for the patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnose with medial osteoarthritis (OA) of the knee with an Alhback score of 2, 3 and 4 (Ahlback 1968) and with any Kujala score for pre-operative anterior knee pain.
* Older than 40 years of age.
* pain on the medial joint line.
* primary medial compartment osteoarthritis with a well preserved lateral compartment with competent cruciate ligaments with correctable intraarticular varus deformity.
* ROM flexion up to 110° under anesthesia.

Exclusion Criteria:

* Patients with fixed varus deformity > 15°
* Inflammatory arthritis
* Previous high tibial osteotomy or ACL reconstruction

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Kujala score | 6 months
  Kujala score including 13 parameters with the score of 0-100, the higher the score the better the function.

SECONDARY OUTCOMES:
complication | 6 months
  number of participant with DVT, infections, loosening of implants, fractures, lateral compartment arthritis, and dislocations of the polyethylene

CONTACTS AND LOCATIONS:
Locations (1):
- Pranungkraw General Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suwankomonkul P, Arirachakaran A, Kongtharvonskul J. Short-term improvement of patellofemoral pain in medial unicompartmental knee arthroplasty with patellar denervation: a prospective comparative study. Musculoskelet Surg. 2022 Mar;106(1):75-82. doi: 10.1007/s12306-020-00675-7. Epub 2020 Aug 2. PMID 32743756